CLINICAL TRIAL: NCT05775354
Title: Reviving Early Diagnosis of Cardiovascular Disease in the Utrecht Health Project
Acronym: RED-LRGP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Monika Hollander, MD, PhD, MD, PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL82944.041.23
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease; Atrial Fibrillation; Heart Failure; Valvular Heart Disease
Keywords: early diagnosis; cardiovascular diseases; cohort study; primary health care
MeSH Terms: conditions — Coronary Artery Disease; Atrial Fibrillation; Heart Failure; Heart Valve Diseases; Disease; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early diagnosis strategy (Experimental): RED-CVD early diagnosis questionnaire, physical examination, laboratory testing, electrocardiography, echocardiography
  Interventions: Diagnostic Test: Early diagnosis strategy
- Usual primary care (No Intervention): No measurements

INTERVENTIONS:
Diagnostic Test: Early diagnosis strategy — RED-CVD early diagnosis questionnaire, physical examination, laboratory testing, electrocardiography, echocardiography
  Arms: Early diagnosis strategy

SUMMARY:
The goal of this randomized trial is to compare the diagnostic yield of a screen-like early diagnosis strategy to usual primary care to detect coronary artery disease (CAD), atrial fibrillation (AF), heart failure (HF), and/or valvular heart disease (VHD) in community people aged 50-80 years who participate in the Utrecht Health Project.

The diagnosis strategy consists of a questionnaire with questions related to symptoms suggestive of CAD, AF or HF, a focused physical examination, laboratory testing, electrocardiography, and echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50-80 years
* Being a participant of LRGP
* Having indicated in the LRGP informed consent to be interested in participating in further research.

Exclusion Criteria:

* Diagnosed with coronary artery disease and atrial fibrillation and heart failure.
* Undergoing major (cardiovascular) surgery, and/or revascularisation therapy and/or transplantation treatment within 3 months after enrolment.
* Not willing to give written informed consent for RED-LRGP.
* Not allowing incidental findings to be reported to him/herself or their own GP.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1476 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Coronary artery disease | 1 year
Atrial fibrillation | 1 year
Heart failure | 1 year
Valvular heart disease | 1 year

SECONDARY OUTCOMES:
Echocardiographic abnormalities | 1 year
Health-related quality of life | 1 year
CVD family history and women's reproductive history | 1 year
Cardiovascular risk profile | 1 year
Costs | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Monika Hollander, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No